CLINICAL TRIAL: NCT04480645
Title: CivaDerm(TM) Surface Therapy Pilot Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: CivaTech Oncology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT008
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Basal Cell Carcinoma; Squamous Cell Carcinoma of the Skin
Keywords: radiation; brachytherapy; skin cancer
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): Radioactive bandage applied to surface of the body worn for approximately one week.
  Interventions: Device: CivaDerm

INTERVENTIONS:
Device: CivaDerm — radioactive bandage

SUMMARY:
This is a pilot study to determine the usefulness of new brachytherapy device that utilizes active components (palladium-103) of standard devices in a novel configuration, which may benefit basal cell and squamous cell carcinoma patients by providing conformal radiation therapy to the surface of the skin.

ELIGIBILITY:
Inclusion Criteria:

* subject signed informed consent
* Confirmed superficial or nodular basal cell or squamous cell carcinoma
* Biopsy proven on chest, stomach, back, arms, legs, feet (trunk and extremities)
* >5 mm of residual tumor
* tumors < 3 cm
* Capable of complying with Patient Release Instructions

Exclusion Criteria:

* Is unable or unwilling to comply with the protocol requirements
* Pregnant or breast feeding
* Metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
skin toxicity events | within 2 months of treatment
  grade 3+ events

SECONDARY OUTCOMES:
dose delivered to target | 1 week
  calculated radiation dose

CONTACTS AND LOCATIONS:
Locations (1):
- CivaDerm Oncology PLLC, Morrisville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No